CLINICAL TRIAL: NCT05863026
Title: Effectiveness of Theory Based Integrated Dengue Education and Learning Module (iDEAL) in Improving the Knowledge, Attitude, Practice, Environmental Cleanliness Index and Dengue Index Among School Children: Study Protocol for a Randomised Controlled Trial
Brief Title: Effectiveness of iDEAL in Improving the Knowledge, Attitude, Practice, Environmental Cleanliness Index and Dengue Index
Acronym: iDEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Takeda Malaysia Sdn. Bhd. (Unknown)
Responsible Party: Principal Investigator, Rahmat bin Dapari, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iDEAL
Record Dates: First submitted 2023-04-25; First posted 2023-05-17 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomised, single blinded, controlled, parallel, trial. This study will recruit and randomise school children into intervention group and control group based on selected school to avoid contamination.
Who Masked: Participant
Masking Description: Allocation concealment In this study, the allocation concealment method that will be use is the "sequentially numbered, opaque, sealed enveloped methods".
  This study will use the single blinding method in which the respondent will not be aware of their group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iDEAL group (Experimental): School cluster randomization will be used to ensure administrative efficacy, lessened risk of experimental contamination, and enhancement of subject compliance. 20 standard 4 classrooms and 20 form 4 classrooms from primary and secondary school, then will be divided randomly into intervention and control group. The unit of randomization will be on a 1:1 basis in either the control or intervention group.
  Interventions: Behavioral: THEORY BASED INTEGRATED DENGUE EDUCATION AND LEARNING MODULE (iDEAL)
- Control (No Intervention): School cluster randomization will be used to ensure administrative efficacy, lessened risk of experimental contamination, and enhancement of subject compliance. 20 standard 4 classrooms and 20 form 4 classrooms from primary and secondary school, then will be divided randomly into intervention and control group. The unit of randomization will be on a 1:1 basis in either the control or intervention group.

INTERVENTIONS:
Behavioral: THEORY BASED INTEGRATED DENGUE EDUCATION AND LEARNING MODULE (iDEAL) — THEORY BASED INTEGRATED DENGUE EDUCATION AND LEARNING MODULE (iDEAL)
  Arms: iDEAL group

SUMMARY:
Background Dengue is a mosquito-borne viral disease caused by four distinct but closely related dengue virus (DENV). The incidence of dengue has grown dramatically worldwide in recent decades, with cases reported to WHO increased from 505,430 cases in 2000 to 5.2 million in 2019. The total number of dengue cases in Malaysia has increased from merely 6,543 cases in the year 1995 to 130,101 cases in the year 2019. Knowledge, attitude and practice remain the most effective driving tool against dengue prevention and control and it becomes very necessary to plan an integrated module for the primary prevention of dengue infection especially among school children.

Aims The present study intends to develop, implement and evaluate the effectiveness of theory-based integrated dengue education module in improving the knowledge, attitude, practice, environmental cleanliness index, and dengue index among school children in Selangor and Kuala Lumpur.

Methods This study is a single-blinded, cluster randomized controlled trial study, expected to be conducted from 1st June 2023 to 31st May 2025 among 20 primary dan 20 secondary schools in Selangor and Kuala Lumpur. The respondents will be allocated into intervention and control groups randomly based on selected clusters to avoid contamination. The intervention group will receive IDEM, while the control group will receive standard education. The outcome will be measured using validated, self-administered questionnaires at four time points: baseline (T0), Immediately (T1), one month (T2), and three months (T3) post-intervention to measure the effectiveness of the intervention module. The data will be analysed using IBM Statistical Package for Social Science (SPSS) version 28 involving descriptive and inferential statistics. The Generalized Linear Mixed Model (GLMM) will be used to test the main effect and interaction between and within the intervention and control groups over time at T0, T1, T2 and T3. This study will use a significance level with a p-value of 0.05 and a confidence interval of 95% for hypothesis testing

DETAILED DESCRIPTION:
Introduction Dengue is a mosquito-borne viral disease caused by four distinct but closely related dengue virus (DENV) serotypes. The incidence of dengue has grown dramatically around the world in recent decades, with cases reported to WHO increased from 505,430 cases in 2000 to 5.2 million in 2019. The total number of dengue cases in Malaysia has increased from merely 6,543 cases in year 1995 to 130,101 cases in year 2019. Knowledge, attitude and behaviour change remain the most effective driving tool against dengue infection and it becomes very necessary to plan an integrated module for primary prevention of dengue infection especially among school children. School-based health education is a crucial tool to enhance knowledge and raise awareness of the seriousness of dengue among school children, and to transfer knowledge and practices from classrooms to homes. The present study intends to develop, implement and evaluate the effectiveness of theory based integrated dengue education module in improving the knowledge, attitude, practice, environmental index and dengue index among school children in Selangor and Kuala Lumpur.

Methods Study design This is a two-arm randomised, single blinded, controlled, parallel, trial.

Study duration The study will be conducted over a period of 24 months, from 1st September 2023 until 31st August 2025, with data collection will be commenced on 1st November 2023.

Study location The study will be conducted in Selangor and Kuala Lumpur.

Study population This study will be carried out in primary and secondary school under supervision of Ministry of Education (MOE). The study participants will be students standard four and form four school children from government primary and secondary school in Selangor and Kuala Lumpur.

Inclusion and exclusion criteria The inclusion criteria for this study are i) Malaysian citizen, ii) standard 4 or form 4 from primary and secondary school respectively, iii) consented to participate in the study by parents or caregivers, and iv) consented by the school. The exclusion criteria i) not able to read Bahasa Malaysia or English, ii) physically or mentally impaired with disability card holder, and iii) temporary student as defined as less than 6 months during the study period.

Sample size estimation The sample size calculation for this study was calculated based on the primary outcome desire which is knowledge on dengue prevention and control. The sample size calculation was calculated using the formula for testing the different in proportion between two groups. After adjustment for attrition rate of 70% from previous study, the sample size needed for this study is 800 pairs of intervention and control groups which amount to 1600 participants.

Sampling method and subject recruitment This study will use a multistage sampling technique. The first stage of sampling will use proportionate sampling base on district in Selangor and Kuala Lumpur to select the 40 schools. One classroom will be selected form each selected school. Thus, the second stage sampling will randomly select 20 standard 4 classrooms and 20 form 4 classrooms from selected primary and secondary school respectively. All school children in selected classroom will be invited to participate in the study.

Randomisation School cluster randomization will be used to ensure administrative efficacy, lessened risk of experimental contamination, and enhancement of subject compliance. 20 standard 4 classrooms and 20 form 4 classrooms from primary and secondary school, then will be divided randomly into intervention and control group. The unit of randomization will be on a 1:1 basis in either the control or intervention group.

Blinding This study will use the single blinding method in which the respondent will not be aware of their group status. This type of blinding aims to minimize performance bias or also known as the Hawthorne effect in which the participant may change their responses or behaviour if they knew which group, they were allocate in (McCambridge et al., 2014). It is not possible to blind the field researcher as they would be the one who will deliver the intervention module to the selected respondents.

Research phase and tools This research protocol details the process of development, implementation, and effectiveness assessment of the theory based integrated dengue education module in improving the knowledge, attitude, practice, environmental cleanliness index and dengue index among school children in Selangor and Kuala Lumpur. The study will be conducted over 24 months, from June 2023 to May 2025. The study consists of three main phases, which are; Phase I: Need assessment Phase II: Development of Intervention module Phase III: Implementation and effectiveness measurement

Phase I: Need assessment Need assessment of the intervention will be conducted through combination approach of community diagnosis. Assessment of the of current knowledge, attitude and practice on dengue prevention and control will be via literature review, survey, Nominal Group Discussion (NGD) and Focus Group Discussion (FGD) among subject matter expert (SME)) and stakeholder. All information will be used for module development (phase II) to design the method and media of delivery, content, and assessment.

Phase II: Development of intervention module A systematic step-by-step procedure will be conducted for designing and developing the Theory Based Integrated Dengue Education Module.

Phase III: Implementation and effectiveness measurement The Implementation of final module will be conducted at selected school. To ensure the standardisation of intervention, trained researcher will conduct the intervention at selected school. To ensure the standardisation, pre-recorded video, briefing and serial supervision by the main investigator will also be practiced throughout the intervention period. Pre and post intervention questionnaire will be collected using validated, self-administered questionnaires at four-time points (T0, T1, T2, T3) to measure the effectiveness of the intervention module.

Questionnaire

A self-administrated questionnaire in two language versions (English and Malay) in printed format will be used in this study. The questionnaire used in the study is a new instrument that will be developed. The questionnaire will be divided into five parts as below:

Part 1: respondent information. Consist of questions of sociodemographic data, socioeconomic and history of dengue infection.

Part 2: Knowledge on dengue prevention and control Part 3: Attitude on dengue prevention and control Part 4: Practice on dengue prevention and control Part 5: Environmental cleanliness index and Aedes index

Validity and reliability Content validity of the questionnaire will be assessed by Subject Matter Experts (SME) that include a public health medicine specialist, family medicine physicians, health educators, occupational health doctor, and occupational-related officer. This evaluation will be performed by various agencies such as the Ministry of Health, NIOSH, DOSH, SOCSO, and Ministry of Higher education. The content validation ratio (CVR) will be calculated to assess the acceptability of the questionnaire. Furthermore, the comments and feedback by the Subject Matter Experts (SME) will be taken into consideration for further correction of the questionnaire. In addition, the Content Validity Index (CVI) will be calculated to assess the relevance and clarity of the questionnaire by the assigned experts. Following that, the Item CVI (I-CVI) and the scale average CVI (S-CVI/Ave) will be calculated. The questionnaire will then be modified according to the agreement level of the experts based on the calculated CVI.

The reliability of the instrument will be measured using internal consistency method calculated in IBM SPSS (Version 28).

Data collection After the initiation of the study, consent will be obtained by the liaison officer from school children who fulfil the eligibility criteria. Subsequently baseline data (T0) will be obtained from school children who consented to join the study. Those subject who consented to join the study and will be allocated in the intervention group will be given appointment within 1 month for delivering of intervention package according to class. The total duration of intervention session will be around 30 minutes for 3 series of meeting. After completion of intervention, the school children will be asked to answer the post intervention assessment measuring outcome of the study immediately (T1), one month (T2) and three months (T3). The control group will undergo the same assessment as the intervention group at baseline, T1, T2 and T3. T

Ethics approval and consent to participate This study has been approved by the Ethics Committee for Research Involving Human Subjects of Universiti Putra Malaysia (JKEUPM-2023-347). All participants will be informed that their enrolment will in no way affect their relationship with their teacher. Consent from each participant parents' or caregiver' will be obtained using a consent form upon agreement to participate in the study before answering the baseline questionnaire. Participants are allowed to withdraw at any point during the study.

Consent for publication and dissemination Consent from the participants for publication will be obtained from the same consent for participation. The results will be reported and presented in international peer-reviewed journals, conferences and other platforms. No personnel or school information will be disclosed in the dissertation writing and other published manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen,
* standard 4 or form 4 from primary and secondary school respectively,
* consented to participate in the study by parents or caregivers,
* consented by the school. The exclusion criteria

Exclusion Criteria:

* not able to read Bahasa Malaysia or English,
* physically or mentally impaired with disability card holder,
* temporary student as defined as less than 6 months during the study period.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
change of knowledge | baseline (T0), immediately post-intervention (T1), one month (T2), and three months (T3) post-intervention
  knowledge score change compare to baseline the unabbreviated scale title: knowledge Score the minimum and maximum values: 15, 75 higher scores mean a better outcome.
change of attitude | baseline (T0), immediately post-intervention (T1), one month (T2), and three months (T3) post-intervention
  attitude score change compare to baseline
  the unabbreviated scale title: Attitude Score the minimum and maximum values: 15, 75 higher scores mean a better outcome.
change of practice | baseline (T0), immediately post-intervention (T1), one month (T2), and three months (T3) post-intervention
  practice score change compare to baseline
  the unabbreviated scale title: Practice Score the minimum and maximum values: 15, 75 higher scores mean a better outcome.

SECONDARY OUTCOMES:
change of Environmental cleanliness index | baseline (T0), immediately post-intervention (T1), one month (T2), and three months (T3) post-intervention
  Environmental cleanliness index score change compare to baseline
  the unabbreviated scale title: Environmental cleanliness index the minimum and maximum values: 3, 15 higher scores mean a better outcome.
change of Aedes index the unabbreviated scale title: Aedes index the minimum and maximum values: 0, 1 higher scores mean a worse outcome. | baseline (T0), immediately post-intervention (T1), one month (T2), and three months (T3) post-intervention
  Aedes index score change compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rahmat Dapari, DrPH, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No